CLINICAL TRIAL: NCT05734417
Title: Effects of Probiotic Against Respiratory & Gastrointestinal Illnesses in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Tze LIONG (Other)
Collaborators: International Islamic University Malaysia (Other); Beijing Scitop Bio-Tech Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIUM-2022-193: UKM-2023-603
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Tract Infections
Keywords: probiotic; respiratory tract infections; Bifidobacterium; children
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Intervention consists of daily administration of excipient plus Bifidobacterium lactis subsp. infantis B8762 at 0.5x10 log colony forming unit (CFU)/day administered daily for 4-weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g/sachet of excipient administered daily for 4-weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral administration of Bifidobacterium lactis subsp. infantis B8762 at 0.5x10 log colony forming unit (CFU)/day for 4-weeks
  Other Names: Bifidobacterium lactis subsp. infantis B8762
  Arms: Probiotic
Dietary Supplement: Placebo — Intervention consists of daily administration of 2g/sachet of excipient administered daily for 4-weeks
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Bifidobacterium lactis subsp. infantis B8762 in treatment of respiratory and gastrointestinal illnesses in children, which are found common among pre-school children in Malaysia aged below 7-years old.

DETAILED DESCRIPTION:
Respiratory and gastrointestinal illnesses are the most common acute diseases in children where no virtually effective treatments or prophylaxes are available for these infections. Probiotics on the other hand have gained increasing evidences as an effective therapy in preventing respiratory and gastrointestinal illnesses. While the precise mechanisms of using probiotics are largely unknown, speculations include: probiotics compete against pathogens; increase the barrier function in respiratory epithelium; immuno-stimulatory effects by enhancing cellular immunity with increased activity of natural killer cells and macrophages in airways and gut. Hence, probiotics may offer safe means of reducing the risk of respiratory and gastrointestinal illnesses, antibiotic use, and the risk of recurrent infections, thereby represent a simple, safe, effective, available and affordable method for preventing respiratory and gastrointestinal infections in children.

Among the various types of probiotics, Bifidobacterium is one of the best-known probiotic genus in the world, and it is widely applied in the dairy industry as a probiotic. Evidences from more than 100 scientific publications based on in vitro, in vivo, and clinical studies and long consumption history support the safety and health benefits of Bifidobacterium strains. The ingestion of yogurt fortified with B. longum reduced harmful bacteria such as Enterobacteriaceae, Streptococcus and C. perfringens, while at the same time alter the microbiota gut profile of volunteers with a significant increase of beneficial microbes Bifidobacterium and Lactobacillus species. Additionally, putrefactive substances in the intestinal environment were also reduced in the presence of the probiotic supplement. Such findings suggest that Bifidobacterium strains are safe and could be used further to evaluate its effect in preventing diarrhea and/or respiratory-related illness prevalence in young children.

Probiotic (Bifidobacterium lactis subsp. infantis B8762) adheres to probiotic properties such as excellent tolerance to gastric acid, intestinal fluid and bile salt of the digestive system. Both probiotic and placebo products are manufactured under an ISO9001, ISO22000 and HACCP conditions. All products do not contain any animal-origin ingredients. The probiotic product contains probiotic and carrier while placebo contains only carrier. Sachets of products containing probiotic and placebo appear as light yellow powder. Both probiotic and placebo products are kept at storage temperature range below 30oC according to the condition recommended by the manufacturer.

A total number of 120 pre-school children with respiratory diseases aged below 7-years old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* preschool children (<7 years old), and having respiratory and/or gastrointestinal diseases symptoms.
* Willing to commit throughout the experiment

Exclusion Criteria:

* Long term medication due to certain severe illness (6 months or more)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 1 Month to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration of respiratory illnesses in children with respiratory tract infections upon administration of probiotic for 4-weeks | 4-weeks
  Changes in duration of respiratory illnesses in children compared between probiotic and placebo after 4-weeks

SECONDARY OUTCOMES:
Clinical respiratory symptoms frequency in children with respiratory tract infections upon administration of probiotic as assessed using the Monthly Health Questionnaire (as used in ClinicalTrials.gov (identifier number NCT02434042). | 4-weeks
  Changes in frequency of respiratory illnesses symptoms from children on probiotic or placebo after 4-weeks, via the use of questionnaire.
Clinical gastrointestinal symptoms in children with respiratory tract infections upon administration of probiotic as assessed using the Monthly Gastrointestinal Questionnaire as used in ClinicalTrials.gov (identifier number NCT02434042). | 4-weeks
  Differences in duration and frequency of gastrointestinal symptoms of children upon administration of probiotic compared to placebo
Microbiota profiles of saliva and fecal samples in children with respiratory tract infections upon administration of probiotic as assessed via pyrosequencing | 4-weeks
  Differences in microbiota abundance of saliva and fecal sample in children with respiratory tract infections upon administration o probiotic compared to placebo
Concentrations of proteins in saliva samples in children with respiratory tract infections upon administration of probiotic as assessed via biochemical tests | 4-weeks
  Differences in concentrations of proteins such as interleukins (IL-10, IL-4, IL-6, Tumour Necrosis Factor-alpha, Interferon gamma) in saliva (ug/mL) samples in children with with respiratory tract infections upon administration of probiotic compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Taufiq Hidayat Hasan, MBBS, Principal Investigator — International Islamic University Malaysia
Locations (1):
- Department of Paediatrics, Kulliyyah of Medicine, IIUM Medical Centre, International Islamic University Malaysia, Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No